CLINICAL TRIAL: NCT06549530
Title: Open-label, Multicenter Immunogenicity and Safety Study of MVA-BN Vaccine in Children From 2 Years to Less Than 12 Years of Age Compared to Adults for the Prevention of Smallpox, Mpox, and Related Orthopoxvirus Infections
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POX-MVA-045
Record Dates: First submitted 2024-07-31; First posted 2024-08-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Monkeypox (Mpox)
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MVA-BN (Experimental): Participants will receive 2 vaccinations at the standard dose of MVA-BN vaccine 4 weeks apart.
  Interventions: Drug: MVA-BN

INTERVENTIONS:
Drug: MVA-BN — All participants will receive 2 vaccinations of the same dose of MVA-BN vaccine 4 weeks apart (standard regimen).

SUMMARY:
All participants will receive 2 vaccinations of the same dose of Modified Vaccinia Ankara Virus (MVA-BN) vaccine 4 weeks apart (standard regimen).

Serum samples for assessment of immune response will be collected at baseline (visit of first vaccination) and at 2 weeks (week 6), 6 months (week 30), and 1 year after the second (last) vaccination.

DETAILED DESCRIPTION:
Both treatment groups will start with enrollment after all study approvals are in place. For the pediatric group, enrollment will open for both age subgroups (children 6 to <12 years of age and 2 to <6 years of age) at the same time. An independent data monitoring committee (DMC) then will review reactogenicity and adverse events (AEs) from both children and adults after at least 10 children in each age subgroup have received the first vaccination and have completed the visit 1 week later. If the DMC assesses the safety data to be positive, the pediatric age subgroups can be opened to full enrollment.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an adult individual must meet all the following criteria:

1. Age 18 to 50 years at screening
2. Male or female sex
3. Informed consent form (ICF) signed and dated by the participant after reading the form and being advised of the risks and benefits of the trial in a language understood by the participant and before performance of any trial-specific procedures
4. General good health, without clinically relevant medical illness, physical exam findings, or laboratory abnormalities, as determined by the investigator
5. Body mass index (BMI) ≥18.5 and ≤35 (calculated as [body weight in kilograms] /[body height in meters] 2)
6. Agreement by female participants of childbearing potential and male participants who are sexually active with a female partner of childbearing potential to use a highly effective method of birth control from at least 30 days prior to administration of the MVA-BN vaccine until 30 days after last vaccination

   1. Medically acceptable methods of contraception that may be used by the participant and/or partner include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone releasing system (IUS), bilateral tubal occlusion, vasectomy, or abstinence (abstinence only acceptable if refraining from heterosexual intercourse during the entire period of 30 days prior to administration of the MVA-BN vaccine until 30 days after last vaccination).
   2. Female participants or partners are not considered to be of childbearing potential if they are at least 1 year post-menopausal (amenorrhea >12 months and follicle stimulating hormone according to local lab values) at screening.
7. Willingness to comply with the requirements of the protocol, in the judgment of the investigator

Pediatric Cohort

To be eligible to participate in this trial, a child must meet all the following criteria:

1. Age ≥2 and <12 years at screening
2. Male or female sex
3. Informed consent form signed and dated by a parent/guardian after reading the form and being advised of the risks and benefits or the trial in a language understood by the parent/guardian and before performance of any trial-specific procedures
4. Assent form signed and dated, for children required by local regulations

   1. provide consent ≥8 years of age enrolled at sites in Uganda
   2. children deemed by the investigator and/or local regulations to be capable of assent in Democratic Republic of Congo
5. General good health, without clinically relevant medical illness, physical exam findings, or laboratory abnormalities, as determined by the investigator
6. Willingness of parent/guardian to comply with the requirements of the protocol, in the judgment of the investigator

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this trial:

1. For female participants: Pregnancy or breastfeeding
2. Acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of responses, including but not limited to, neurologic, cardiovascular, respiratory, hepatic, hematologic, rheumatologic, endocrine, gastrointestinal, renal, autoimmune, or immunosuppressive conditions
3. History of or active autoimmune disease (vitiligo or thyroid disease requiring thyroid replacement are not exclusions), history of Guillain-Barré syndrome or Reye's syndrome
4. Known immunodeficiency syndrome or known or suspected impairment of immunologic functions including, but not limited to, clinically significant liver disease, diabetes mellitus type I, or moderate to severe kidney impairment. Human immunodeficiency virus (HIV) infection under stable Highly active antiretroviral therapy (HAART) (no change within the last three month) and CD4 count >500/ µL is not considered immunodeficient
5. Known or reported previous smallpox vaccination, or vaccination with any licensed or investigational poxvirus-based vaccine
6. History of monkeypox, cowpox, or vaccinia infection
7. Close contact in the 3 weeks prior to signing the ICF with anyone known to have mpox
8. History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months prior to screening that is considered to have achieved cure
9. Clinically significant mental disorder not adequately controlled by medical treatment
10. Active or recent (within 6 months before screening) chronic alcohol abuse and/or intravenous and/or nasal drug abuse
11. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, eg, tris(hydroxymethyl)-amino methane, including history of allergic asthma
12. Known allergy to aminoglycosides or quinolones
13. History of anaphylaxis of severe allergic reaction to any vaccine
14. Receipt of or plans to receive any licensed live vaccine from 30 days prior to the trial vaccination until 30 days after vaccination
15. Receipt of or plans to receive any licensed nonlive vaccine from 14 days prior to the trial vaccination until 14 days after last trial vaccination
16. Use of any investigational or nonregistered agent within 30 days prior to vaccination or plans to receive an investigational agent during the trial
17. Recent blood donation (including platelets, plasma, and red blood cells) within 4 weeks prior to screening or planned blood donations during the active trial period
18. Chronic systemic administration (defined as more than 14 days) of >5 mg prednisone (or equivalent)/day or any other immune-modifying drugs from 3 months prior to the first trial vaccination to the visit at the end of the active trial period (use of topical, inhaled, ophthalmic, and nasal glucocorticoids is allowed)
19. History of organ transplantation, whether or not chronic immunosuppressive therapy. is being administered
20. Administration or planned administration of immunoglobulins and/or any blood products from 3 months prior to the first trial vaccination until the visit at the end of the active trial period (packed red blood cells given for an emergency indication in an otherwise healthy person and not required as ongoing treatment is not exclusionary [eg, packed red blood cells given in an emergency during elective surgery])
21. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, significant arrhythmia with or without corrective/ablative surgery, or any other heart condition under the care of a doctor
22. Employment with the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or relationship to the investigator or study site employee
23. Relationship with Bavarian Nordic as an employee or employee family member, contractor, agent, or business partner or a financial interest in the outcome of the trial

Pediatric Cohort

A child who meets any of the following criteria will be excluded from participation in this trial:

1. Acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of responses, including but not limited to, neurologic, cardiovascular, respiratory, hepatic, hematologic, rheumatologic, endocrine, gastrointestinal, renal, autoimmune, or immunosuppressive conditions
2. History of or currently active autoimmune disease (vitiligo or thyroid disease requiring thyroid replacement therapy are not exclusions), history of Guillain-Barré syndrome or Reye's syndrome
3. Known immunodeficiency syndrome. or known or suspected impairment of immunologic functions including, but not limited to, clinically significant liver disease, diabetes mellitus type I, or moderate to severe kidney impairment. HIV infection under stable HAART (no change within the last three month) and CD4 count >500/ µL is not considered immunodeficient
4. Known or reported previous smallpox vaccination or vaccination with any licensed or investigational poxvirus-based vaccine
5. History of monkeypox, cowpox, or vaccina infection
6. Close contact in the 3 weeks prior to signing the ICF/assent form with anyone known to have mpox
7. History of malignancy (eg, leukemia or lymphoma)
8. History of chronic or known neurological disease or deficient development history
9. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including history of allergic asthma
10. Known allergy to aminoglycosides or quinolones
11. History of anaphylaxis or severe allergic reaction to any vaccine
12. Receipt of or plans to receive any licensed live vaccine from 30 days prior to first trial vaccination until 30 days after last trial vaccination
13. Receipt of or plans to receive any licensed nonlive vaccine from 14 days prior to first trial vaccination until 14 days after last trial vaccination
14. Use of any investigational or nonregistered agent other than the trial vaccine within 30 days prior to first vaccination or plans to receive an investigational agent during the trial period
15. Chronic administration (defined as more than 14 days) of systemic high dose immune suppressant drugs (2 mg/kg/day or more of prednisolone or its equivalent or 20 mg/day or more for children who weigh more than 10 kg) from 6 months prior to first trial vaccination to trial conclusion
16. History of organ transplantation, whether or not chronic immunosuppressive therapy. is being administered
17. Administration or planned administration of immunoglobulins and/or any blood products from 3 months prior to the first trial vaccination until the visit at the end of the active trial period
18. Employment of parent/guardian with the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or relationship to the investigator or study site employee
19. Relationship of parent/guardian with Bavarian Nordic as an employee or employee family member, contractor, agent, or business partner or a financial interest in the outcome of the trial

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of 2 doses of MVA BN | 2 weeks after the second MVA-BN vaccination
  Titer of serum neutralizing antibodies against vaccinia virus as measured by plaque reduction neutralization tests (PRNTs) 2 weeks after the second MVA BN vaccination
Occurrence of Safety Adverse Events (SAE) & Adverse of Event of Special Interest (AESI) events | Day 0 to week 56
  Occurrence of any SAE at any time during the trial period Occurrence of any AESI at any time during the trial period

SECONDARY OUTCOMES:
Neutralizing antibody response | From day zero to two weeks after the second vaccination
  To assess neutralizing antibody response to the MVABN standard regimen
Neutralizing antibody response durability | Six months and one year after the second vaccination
  To assess durability of neutralizing antibody response to the MVABN standard regimen

CONTACTS AND LOCATIONS:
Locations (3):
- University of Kinshasa, Kinshasa, Democratic Republic of the Congo
- Uganda (2):
  - Uganda Virus Research Institute, Entebbe
  - Epicentre Mbarara Research Centre, Mbarara

IPD SHARING:
Plan to Share IPD: No